CLINICAL TRIAL: NCT03936751
Title: Impact of Obstructive Sleep Apnea Treatment on Cardiovascular Events in Patients With Acute Cardiogenic Pulmonary Edema: a Multicenter Randomized Controlled Study (CPAP-CARE STUDY).
Brief Title: Obstructive Sleep Apnea Treatment on Cardiovascular Events in Patients With Acute Cardiogenic Pulmonary Edema: CPAP-CARE STUDY.
Acronym: CPAP-CARE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID-19 pandemic and philips cpap machine recall
Sponsor: University of Sao Paulo (Other)
Collaborators: Philips Respironics (Industry); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Luciano F Drager, MD, PhD, Associate Professor of Medicine, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SDC 4782/18/148
Record Dates: First submitted 2019-04-05; First posted 2019-05-03 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Obstructive Sleep Apnea; Pulmonary Edema Cardiac Cause
MeSH Terms: conditions — Sleep Apnea, Obstructive; Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CPAP (Active Comparator): Continuous positive airway pressure
  Interventions: Device: CPAP
- Nasal strips (Sham Comparator): Nasal Strips
  Interventions: Device: Nasal Strips

INTERVENTIONS:
Device: CPAP — This is the standard treatment for OSA.
  Arms: CPAP
Device: Nasal Strips — Nasal strips were commercially available in the market for supposing treat snoring and sleep apnea but no proof that this is true. Our group previously validated nasal strips as an interesting placebo.
  Arms: Nasal strips

SUMMARY:
Despite the advances in the treatment of acute cardiogenic pulmonary edema (ACPE), the readmissions rates and cardiovascular events remain very high. In this context, it is possible that other potential risk factors may influence the poor prognosis of the ACPE. One of these potential candidates is Obstructive Sleep Apnea(OSA). This study was designed to evaluate the impact of OSA treatment with CPAP in consecutive patients with ACPE. The primary outcome will be to evaluate the impact of CPAP on the recurrence of ACPE in the 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive acute Cardiogenic Pulmonary Edema
* Moderate to Severe OSA

Exclusion Criteria:

* Professional drivers
* Pregnancy
* Non-Cardiogenic Pulmonary edema
* Terminal cancer

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of ACPE recurrence | 1-year
  To evaluate the effects of CPAP on the recurrence of ACPE as compared to placebo

SECONDARY OUTCOMES:
Rate of all-cause mortality | 1-year
  To evaluate the effects of CPAP on the all-cause mortality as compared to placebo
Rate of cardiovascular mortality | 1-year
  To evaluate the effects of CPAP on the cardiovascular mortality as compared to placebo
Number of new hospital admissions | 1-year
  To evaluate the effects of CPAP on the number of new hospital admissions as compared to placebo
Blood pressure effects ( (mmHg) | 1-year
  To evaluate the effects of CPAP on the blood pressure reduction as compared to placebo
Levels of BNP levels (pg/ml) | 1-year
  To evaluate the effects of CPAP on the BNP levels as compared to placebo
Cardiac function (left ventricular ejection fraction - %) | 1-year
  To evaluate the effects of CPAP on the left ventricular ejection fraction (by echocardiography) as compared to placebo

CONTACTS AND LOCATIONS:
Locations (4):
- Brazil (4):
  - PROCAPE - University of Pernambuco, Recife, São Paulo
  - Hospital Samaritano, São Paulo, São Paulo
  - Heart Institute (InCor), São Paulo
  - Hospital Dante Pazzanese, São Paulo

IPD SHARING:
Plan to Share IPD: No